CLINICAL TRIAL: NCT01722955
Title: Effect of Pre-warmed Intravenous Fluids on the Early Outcomes After Ambulatory Surgery Under Monitored Anesthesia Care
Brief Title: Pre-warmed Intravenous Fluids and Monitored Anesthesia Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung Hee Kim, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Prewarmed fluid
Record Dates: First submitted 2012-11-04; First posted 2012-11-07 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Hypothermia
Keywords: Prewarmed fluid; monitored anesthesia care; core body temperature; anesthetic satisfaction
MeSH Terms: conditions — Hypothermia | interventions — Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-warmed fluids (Experimental): Pre-warmed fluids will be prepared for 8hous in 41℃ set hot cabinet.
  Interventions: Other: Pre-warmed fluids
- Room temperature fluids (Experimental): Room temperature fluids will be stored at ambient temperature.
  Interventions: Other: Room temperature fluids

INTERVENTIONS:
Other: Pre-warmed fluids — IV fluid will be stored at 41℃ set hot cabinet for 8hours
  Other Names: Warming intravenous (IV) fluid
  Arms: Pre-warmed fluids
Other: Room temperature fluids — Room temperature fluid will be stored at ambient temperature
  Other Names: No warming intravenous fluids
  Arms: Room temperature fluids

SUMMARY:
The aim of the study is to compare effect of pre-warmed intravenous fluids on the early outcomes in ambulatory patients undergoing monitored anesthesia care.

DETAILED DESCRIPTION:
Monitored anesthesia care (MAC) has been increasing in fast track anesthesia for ambulatory or outpatient surgery. MAC provides lower anesthetic agents than general anesthesia, however it has been shown to result high anesthetic complication rate because of negligent monitoring. Therefore, aim of this study is to investigate the effect of pre-warmed intravenous fluids on the core body temperature and the early outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 20years to 70years old female patients undergoing urinary incontinence surgery under monitored anesthesia care.

Exclusion Criteria:

* Preoperative tympanic membrane temperature >38 or < 36
* End stage heart failure or renal failure
* Otitis media

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Tympanic membrane temperature | 30min after anesthetic induction
  Preoperative dehydration will be supplemented with 10ml/kg of lactate Ringer's solution at the beginning of the anesthetic induction. 30 min after anesthetic induction is nearly after administering the fixed volume.

SECONDARY OUTCOMES:
Postoperative chilling and shivering | on arrival at the postanesthetic care unit ( 1hour after the anesthetic induction)
  Degree of chilling and shivering will be evaluated at the postanesthesia care unit after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Myung Hee Kim, MD,PhD, Principal Investigator — Samsung MC
Locations (1):
- Samsung medical center, Seoul, South Korea

REFERENCES:
- [Result] Yokoyama K, Suzuki M, Shimada Y, Matsushima T, Bito H, Sakamoto A. Effect of administration of pre-warmed intravenous fluids on the frequency of hypothermia following spinal anesthesia for Cesarean delivery. J Clin Anesth. 2009 Jun;21(4):242-8. doi: 10.1016/j.jclinane.2008.12.010. Epub 2009 Jun 6. PMID 19502035